CLINICAL TRIAL: NCT07009028
Title: The Effect of Storigami Method on Pain, Fear and Anxiety Levels Associated With Peripheral Intravenous Catheterisation in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Ayşe Kahraman, Assoc. Prof. Dr., Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 125S582
Record Dates: First submitted 2025-05-20; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Pain
Keywords: nurse; child; distraction methods
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: The population of the randomized controlled experimental study consisted of children aged 6-9 years who were admitted to the Pediatrics Clinic and hospitalized in the hospital.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arms (No Intervention): No Intervention: children will receive standard care during peripheral intravenous catheterization.
- Arm (Experimental): Experimental:storigami method will be applied during peripheral intravenous catheterization of children
  Interventions: Combination Product: Storigami figure

INTERVENTIONS:
Combination Product: Storigami figure — Combination Produc: The origami figure that will be formed as a result of the process will be used as a distraction method
  Arms: Arm

SUMMARY:
The aim of this study was to determine the effect of storigami method on reducing pain, fear and anxiety of children in peripheral intravenous catheter applications in children aged 6-9 years who were hospitalized in the pediatric health and diseases clinic.

DETAILED DESCRIPTION:
He stated that children and their families who frequently visit hospitals for follow-up, treatment or various anomalies have negative hospital experiences due to fear, anxiety and painful procedures, and that these negative experiences may cause phobias and avoidance of medical procedures in children in the future. Therefore, this study was planned to determine the effect of storigami method on reducing pain, fear and anxiety of children in peripheral intravenous catheter applications in children aged 6-9 years who were hospitalized in the pediatric health and diseases clinic. Storigami is a method that involves the use of origami and stories at the same time and can be used to reduce pain in hospitals. The method, which is planned to be used to minimize negative hospital experiences, is thought to be a promising, cost-effective and safe non-pharmacological technique that can be used safely to reduce fear, anxiety and pain of hospitalized patients.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* The child is between 6-9 years old
* First time peripheral intravenous catheter insertion since admission to the clinic
* The child has no vision, hearing and speech problems
* The child has no mental retardation
* Know/speak Turkish
* No complaints such as pain, nausea and vomiting that may affect fear and anxiety
* No sedative or analgesic was given to the child immediately before the peripheral intravenous catheterization procedure

Exclusion Criteria:

* The child has a chronic, congenital, metabolic or neurodegenerative disease
* Failed attempt at peripheral intravenous catheterization,
* Failure to complete or incomplete completion of questionnaires,
* A different invasive intervention was performed immediately before PIC application,
* The child does not comply during the procedure,
* The child wants to leave the study

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-08-20 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Reducing the child's fear | during peripheral intravenous procedure
  The Children's Fear Scale (CFS) was graded on a scale of 0-4 and included five display images with facial expressions ranging from neutral (0 = no anxiety) to fearful (4 = severe anxiety). Children between the ages of 5 and 10 can use it before and after treatments.
  For child and proxy reports, it contain different instructions to reduce the child's fear during the peripheral intravenous catheterization procedure.
Reducing the child's anxiety | during peripheral intravenous procedure
  Child Anxiety Scale-State (CASsingle bondS). Its bottom resembles a lightbulb, and its horizontal lines with upward ranges like those of a thermometer. To measure state anxiety, the child is asked to say that he feels "now" It applied to kids ages 4 to 12 and had a range of 0 to 10. There is a direction in the scale "NOW color where you FEEL on the thermometer, too much tension or anxious, calm: not tension or anxious? Children were asked to "Pretend that all your worried or nervous feelings are in the very bottom down here (point to scale). If you are a little bit worried or nervous, the feelings might come up just a little bit (move your finger up). If you are very, very worried or nervous, the feelings might go all the way to the top (move your finger up to the top). Put a line showing how much worry or nervousness you feel." It ranges from 0 to 10 and can be applied to children aged 4-12.
  Reduce the child's anxiety during the peripheral intravenous catheterization procedure
Reducing the child's pain | during peripheral intravenous procedure
  This scale, which has six faceted expressions and assigns a pain score based on the numerical values of the faces, is used to diagnose pain in children. It is used to assess the pain in children three years and older. Faces can display a range of emotions, from crying (10 = most painful) to smiling (0 = no pain)
  reduce the child's pain during the peripheral intravenous catheterization procedure

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Kahraman, Assoc Prof, Principal Investigator — Ege Universty
Locations (2):
- Turkey (Türkiye) (2):
  - Ege University, Izmir, Bornova
  - Ege University, Izmir, İzmir

IPD SHARING:
Plan to Share IPD: No